CLINICAL TRIAL: NCT00002824
Title: A PHASE I TRIAL OF HSV-TK ADENOVIRUS GENE THERAPY FOR PRIMARY BRAIN TUMORS
Brief Title: Gene Therapy in Treating Patients With Primary Brain Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065004; UPCC-3394; NCI-H96-0976
Record Dates: First submitted 1999-11-01; First posted 2004-07-29 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2000-07

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Gliosarcoma | interventions — Genetic Therapy; Drug Therapy; Ganciclovir

INTERVENTIONS:
Biological: gene therapy
Drug: chemotherapy
Drug: ganciclovir
Procedure: conventional surgery

SUMMARY:
RATIONALE: Inserting the gene for herpes virus into a person's cells may improve the body's ability to fight cancer or make the cancer more sensitive to chemotherapy using antiviral drugs such as ganciclovir.

PURPOSE: Phase I trial to study the effectivenesss of gene therapy in treating patients with primary brain tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the response to a stereotactically administered recombinant adenovirus vector carrying the herpes simplex virus thymidine kinase gene (H5.010RSVTK) followed by intravenous ganciclovir in patients with recurrent malignant glioma. II. Estimate the maximum tolerated dose of H5.010RSVTK in these patients. III. Describe the toxic effects of H5.010RSVTK. IV. Assess the efficiency of gene transfer and duration of transgene expression in these patients. V. Assess quantitative and qualitative glucose metabolic activity of tumoral sites by positron emission tomography. VI. Analyze the immunologic response to adenovirus transduction in these patients. VII. Determine the benefit and toxicity of multiple doses of H5.010RSVTK in patients with resectable tumors.

OUTLINE: This is a dose-finding study. All patients receive stereotactically injected H5.010RSVTK (a recombinant adenovirus vector containing the herpes simplex virus thymidine kinase gene). Cohorts of 3-6 patients receive escalating doses of H5.010RSVTK until the maximum tolerated dose is reached. Ganciclovir is then given on the third post-injection day. Patients with unresectable tumors receive ganciclovir for 14 consecutive days. Patients with resectable tumors receive ganciclovir for 7 consecutive days before undergoing craniotomy with optimal debulking and injection of a second dose of the adenovirus vector followed by ganciclovir for 14 more days. Patients are followed monthly for survival.

PROJECTED ACCRUAL: A total of 18 patients (9 with resectable tumors and 9 with unresectable tumors) will be entered over 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed malignant glioma, including: Anaplastic astrocytoma Glioblastoma Evidence of recurrence by MRI and positron emission tomography despite primary treatment that included radiotherapy with or without chemotherapy Stereotactically accessible tumor Solitary tumor preferred Largest tumor surgically accessible for debulking if multifocal disease Not adjacent to optic chiasm or brain stem No subependymal spread No herniation or marked midline shift Consent for autopsy required

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70%-100% Hematopoietic: Hematologic parameters normal Hepatic: Hepatic parameters normal (less than twice normal if on anticonvulsants) Renal: Renal parameters normal Cardiovascular: No congestive heart failure No angina Other: No medical contraindication to neurosurgery and fluid injection into brain No serious uncontrolled infection Negative pregnancy test required of fertile women prior to entry Adequate contraception required of fertile women during and for 3 months after treatment

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics At least 2 months since radiotherapy Surgery: Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1996-02

CONTACTS AND LOCATIONS:
Overall Officials: Jane B. Alavi, MD, Study Chair — Abramson Cancer Center at Penn Medicine
Locations (1):
- University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania, United States